CLINICAL TRIAL: NCT05059327
Title: A Phase 2B, Multicenter, 30-week, Prospective, Cross-over, Double-blind, Randomized, Placebo-controlled Study Followed by a 52-Week Open-label Extension Study to Evaluate the Efficacy and Safety of Basimglurant Adjunctive to Ongoing Anticonvulsive Therapy in Children, Adolescents, and Young Adults With Uncontrolled Seizures Associated With Tuberous Sclerosis Complex
Brief Title: Basimglurant (NOE-101) in Children, Adolescents, and Young Adults With TSC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Noema Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NOE-TSC-201
Record Dates: First submitted 2021-08-20; First posted 2021-09-28 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Tuberous Sclerosis Complex
Keywords: Basimglurant; TSC; Seizures; NOE-101
MeSH Terms: conditions — Tuberous Sclerosis; Seizures | interventions — 2-chloro-4-(1-(4-fluorophenyl)-2,5-dimethyl-1H-imidazol-4-ylethynyl)pyridine

STUDY DESIGN:
Intervention Model Description: This is a multi-center, randomized, double-blind, placebo-controlled, 30-week, cross-over (Part A) followed by a 52-week open-label extension (OLE) (Part B) study.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Basimglurant/NOE-101 to Placebo) (Experimental): Basimglurant to Placebo
  Interventions: Drug: Basimglurant with crossover to Placebo
- Arm B (Placebo to Basimglurant/NOE-101) (Placebo Comparator): Placebo to Basimglurant
  Interventions: Drug: Placebo with crossover to Basimglurant

INTERVENTIONS:
Drug: Basimglurant with crossover to Placebo — Basimglurant with crossover to Placebo
  Arms: Arm A (Basimglurant/NOE-101 to Placebo)
Drug: Placebo with crossover to Basimglurant — Placebo with crossover to Basimglurant
  Arms: Arm B (Placebo to Basimglurant/NOE-101)

SUMMARY:
The study intends to show that basimglurant (NOE-101) provides effective seizure control in children, adolescents and young adults with Tuberous Sclerosis Complex (TSC).

DETAILED DESCRIPTION:
The study drug (NOE-101, basimglurant) is a potent inhibitor of metabotropic glutamate receptor 5 (mGluR5) which controls a wide range of processes in the brain, spinal cord, retina, and peripheral nervous system. In animal studies, the inhibition of this receptor has shown therapeutic potential for the treatment of Tuberous Sclerosis Complex (TSC). This receptor's inhibition decreases the frequency of seizures. In previous clinical trials, the study drug has shown an advantageous safety profile in children and adolescents.

The objective of this study is to find an optimal dose at which the study drug will lead to a decrease in the duration, frequency and intensity of seizures in children, adolescents and young adults with TSC, while being well tolerated. All patients who positively respond and tolerate the medicine will be offered the possibility to continue in an open label extension.

ELIGIBILITY:
Inclusion Criteria (summary):

* Ability and willingness to provide informed assent or written consent or consent from their legal representative.
* Fluency in the language of the study staff
* Age 5 to 30 years at study entry
* A documented history of TSC
* Refractory seizure history
* Currently receiving one or more anti-epileptic drugs (AEDs)
* Stable medications or interventions for epilepsy
* Willingness to complete Patient Reported Outcome assessments
* For female patients of childbearing potential:

  1. Willingness to undergo serum or urinary pregnancy testing at screening and during the trial period.
  2. Willingness to use contraception.

Exclusion Criteria (summary):

* Neurologic disease other than TSC
* Recent anoxic episode
* Patient weight below 15kg
* Clinically significant unstable medical condition(s)
* Pregnancy or lactation

Ages: 5 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Mean percentage in monthly seizure frequency during the maintenance dosing in Period 2 (Weeks 13 to 16) and Period 4 (Weeks 27-30). | 30 weeks

SECONDARY OUTCOMES:
Number of patients considered treatment responders. | 30 weeks
Longest seizure free interval (i.e., seizure free days). | 30 weeks
Change in the severity of symptoms of TSC as measured by Caregiver Global Impression of Change (CGIC) score during maintenance dosing in Period 2 (Weeks 13 to 16) and Period 4 (Weeks 27-30) compared to Baseline. | 30 weeks
Change in the Sheehan Disability Scale during maintenance dosing in Period 2 (Weeks 13 to 16) and Period 4 (Weeks 27-30) compared to baseline. | 30 weeks
Safety of the study drug in children, adolescents and young adults with seizures associated with TSC. | 82 weeks
  Measured in terms of incidence, nature, and severity of adverse events, vital signs, physical examination, clinical chemistry, hematology, electrocardiograms, and urinalysis, as well as treatment delays, dose reductions, and dose discontinuations. In addition, suicidal ideation will be assessed using S-STS.

OTHER OUTCOMES:
Change in seriousness of disease as assessed by Most Impactful Symptoms Scale in Periods 2 (weeks 13 to 16) and Period 4 (weeks 27 to 30) compared to baseline. | 30 weeks
Frequency of seizures detected by the wearable device evaluated as the change from Baseline compared to study treatment in Period 1 (weeks 13 to 16) and Period 4 (weeks 27 to 30). | 30 weeks
Intensity of seizures detected by the wearable device evaluated as the change from Baseline compared to study treatment Periods 1 and 4. | 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Director, MD, Study Director — Noema Pharma AG
Locations (27):
- United States (9):
  - David Geffen School of Medicine at UCLA (Site #: 101), Los Angeles, California
  - Kennedy Krieger Institute (Site #: 110), Baltimore, Maryland
  - Boston Children's Hospital (Site #: 102), Boston, Massachusetts
  - William Beaumont Hospital - Royal Oak (Site #: 104), Royal Oak, Michigan
  - Minnesota Epilepsy Group PA (Site #: 105), Roseville, Minnesota
  - Boston Children's Health Physicians (BCHP) (Site #: 111), Hawthorne, New York
  - Duke Children's Hospital and Health Center (Site #: 106), Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Rainbow Babies and Childrens Hospital (Site #: 107), Cleveland, Ohio
  - The University of Texas Medical School at Houston (Site #: 103), Houston, Texas
- India (6):
  - Citi Neuro Centre (Site # 806), Hyderabad, Andhra Pradesh
  - Rainbow Childrens Hospital (Site # 803), Hyderabad, Andhra Pradesh
  - Jaslok Hospital and Research Centre (Site # 801), Mumbai, Maharashtra
  - Deenanath Mangeshkar Hospital and Research Centre (Site # 805), Pune, Maharashtra
  - All India Institute of Medical Sciences (Site # 804), New Delhi, National Capital Territory of Delhi
  - Christian Medical College (Site # 807), Vellore, Tamil Nadu
- Hadassah Medical Center - PPDS (Site #: 503), Jerusalem, Israel
- ASST Grande Ospedale Metropolitano Niguarda - Presidio Ospedaliero Ospedale Niguarda (Site # 183), Milan, Lombardy, Italy
- Instytut Pomnik Centrum Zdrowia Dziecka (Site # 262), Warsaw, Masovian Voivodeship, Poland
- Spain (4):
  - Hospital Universitario Germans Trias i Pujol (Site # 194), Badalona, Barcelona
  - Hospital Sant Joan de Deu - PIN (Site # 192), Esplugues de Llobregat, Barcelona
  - Hospital Regional Universitario de Malaga - Hospital General (Site # 193), Málaga
  - Centro de Neurología Avanzada (Site # 191), Seville
- Turkey (Türkiye) (3):
  - Istanbul Universitesi Istanbul Tip Fakultesi Hastanesi (Site #: 905), Fatih, Istanbul
  - Yeditepe University Kosuyolu Hospital (Site #: 904), Kadıköy, Istanbul
  - Istanbul Egitim ve Arastirma Hastanesi (Site #: 901), Sultangazi, Istanbul
- United Kingdom (2):
  - Salford Royal Hospital - PPDS (Site # 304), Salford, Lancashire
  - Noahs Ark Children's Hospital (Site # 306), Cardiff, South Glamorgan